CLINICAL TRIAL: NCT01587170
Title: Phase 2: Effects of Zolmitriptan on Sensory Afferent Transmission After Spinal Cord Injury
Brief Title: Effects of Zolmitriptan on Sensory Transmission After Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00019967
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Spinal Cord Injuries; Muscle Spasticity
Keywords: spasticity; spinal cord injury; zolmitriptan
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity

GROUPS / COHORTS (2):
- Uninjured control subjects: Uninjured, control subjects who are not taking any of the contraindicated drugs.
- Spinal-cord injured subjects: Patients who have suffered a spinal cord injury (>1year ago).

SUMMARY:
After spinal cord injury, patients develop a spastic syndrome that is characterized by hyperactive reflexes, increased muscle tone, clonus and involuntary muscle spasms. The neuronal mechanisms behind the development of spasticity remain largely unknown, though animal experiments have shown that changes occur both at the level of the motoneuron and sensory neurons. This project aims to examine the changes that occur in the modulation of sensory afferent transmission after spinal cord injury, and how these changes can contribute to the triggering and initiation of muscle spasms after chronic spinal cord injury in humans.

It is known that after spinal cord injury, the majority of descending sources of monoamines, such as serotonin (5HT), are abolished. Animal experiments have shown that 5HT receptors on sensory neurons in the spinal cord are responsible for inhibiting sensory transmission. As a result, after spinal cord injury these receptors are no longer activated below an injury, resulting in the production of large, long excitatory responses in the motoneuron when sensory are activated. This large sensory activation of the motoneuron can, in turn, activate a long response in the motoneuron to produce an involuntary muscle spasm. The aim of our study is to determine whether, similar to animal experiments, the 5HT1 receptors are responsible for sensory inhibition in spinal cord injured subjects, and whether activating these receptors (through the 5HT1 agonist Zolmitriptan) will restore the normal inhibition of sensory transmission that is lost after injury, thereby resulting in a decrease in the initiation of involuntary muscle spasms.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have suffered a trauma to the spinal cord at least 1 year prior. In addition, subjects must exhibit some degree of spasticity as determined by having an Ashworth Spasticity Score greater than 1 in the ankle or knee.

Exclusion Criteria:

* If patients have damage to the nervous system other than to the spinal cord
* Pregnant women
* Elderly Patients (> 65 years)
* Alcoholic Patients
* History of ischemic cardiac, cerebrovascular or peripheral vascular syndromes
* Valvular heart disease or cardiac arrhythmias
* Other significant underlying cardiovascular disease (atherosclerotic disease, congenital heart disease)
* Uncontrolled or severe hypertension
* Hemiplegic, basilar or ophthalmologic migraine
* Hypersensitivity to Zolmitriptan or any component of the formulation
* History of Autonomic Dysreflexia
* Patients taking:
* Ergot-containing drugs
* Other 5HT1 Agonists
* MAO Inhibitors
* Cimetidine and other 1A2 Inhibitors
* Propranolol
* Selective Serotonin and Norepinephrine Reuptake Inhibitors
* Acetaminophen
* Metoclopramide
* Xylometazoline
* Oral Contraceptives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Spinal cord injury subjects
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in H-reflex amplitude from baseline | Pre baseline, 30, 60, 90 and 120 minutes
  H-reflexes in the soleus muscle will be evoked by stimulation of the posterior tibial nerve. The response will recorded before drug intake, and every 30 minutes after drug intake up to 2 hours to determine the change in the response as a result of drug intake.
Change in Cutaneomuscular Reflex Responses from baseline | Pre baseline, 30, 60, 90, 120 minutes
  Tibialis anterior reflex responses will be recorded after medial arch stimulation of the foot. Recordings will be taken to provide a pre-drug baseline and then every 30 minutes after drug intake up to 2 hrs to determine the change in these reflex responses after drug intake.

SECONDARY OUTCOMES:
Change in Blood pressure | Pre and 60min, 120min post drug
  Blood pressure will be measured to determine the safety of the drug during the study.
Change in Heart rate | Predrug, 60min and 120min after drug
  Heart rate will be monitored before drug intake and 60 and 120 min after drug intake so as to monitor vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Gorassini, PhD, Principal Investigator — University of Alberta; Ming Chan, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Murray KC, Stephens MJ, Rank M, D'Amico J, Gorassini MA, Bennett DJ. Polysynaptic excitatory postsynaptic potentials that trigger spasms after spinal cord injury in rats are inhibited by 5-HT1B and 5-HT1F receptors. J Neurophysiol. 2011 Aug;106(2):925-43. doi: 10.1152/jn.01011.2010. Epub 2011 Jun 8. PMID 21653728
- See also: Related Info — http://www.scialberta.ca/